CLINICAL TRIAL: NCT00257998
Title: Comparison of the Effectiveness of Three Manual Physical Therapy Techniques in a Subgroup of Patients With Low Back Pain Who Satisfy a Clinical Prediction Rule: A Randomized Clinical Trial.
Brief Title: Effectiveness of Three Manual Physical Therapy Techniques in a Subgroup of Patients With Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Franklin Pierce University (Other)
Collaborators: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIC 05-17
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Procedure: Mobilization — manualtherapy techniques

SUMMARY:
Recently a clinical prediction rule (CPR) has been developed and validated that accurately identifies patients with low back pain that are likely to benefit from a lumbo-pelvic manipulation. The studies that developed and validated the rule used the identical manipulation procedure. However, recent evidence suggests that different manual therapy techniques may result in the same outcome.Purpose: The purpose of this study is to investigate the effectiveness of three different manual therapy techniques in a subgroup of patient with low back pain that satisfy the CPR.

ELIGIBILITY:
Inclusion Criteria:

1. Chief complaint of pain and/or numbness in the lumbar spine, buttock, and/or lower extremity
2. Oswestry disability score of at least 25%
3. Age greater than 18 years and less than 60 years
4. At least four out of five of the following criteria:

   1. Duration of current episode < 16 days (judged from the patient's self-report)
   2. No symptoms extending distal to the knee (judged from the pain diagram)
   3. FABQ-W score <19
   4. At least one hip with >350 internal rotation range of motion (measured in prone)
   5. Stiffness in the lumbar spine (judged from segmental mobility testing)

Exclusion Criteria:

1. Red flags noted in the participant's general medical screening questionnaire (i.e. tumor, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, etc.)
2. Signs consistent with nerve root compression, this includes any one of the following:

   1. Reproduction of low back or leg pain with straight leg raise at less than 450
   2. Muscle weakness involving a major muscle group of the lower extremity
   3. Diminished lower extremity muscle stretch reflex (Quadriceps or Achilles tendon)
   4. Diminished or absent sensation to pinprick in any lower extremity dermatome
3. Prior surgery to the lumbar spine or buttock
4. Current pregnancy
5. Past medical history of osteoporosis or spinal compression fracture
6. Inability to comply with treatment schedule (weekly sessions for four weeks)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The Oswestry Disability Index, which will serve as the primary outcome measure. | 4 weeks, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Cleland, DPT, OCS, Principal Investigator — Franklin Pierce University
Locations (1):
- Rehabilitation Services of Concord Hospital, Concord, New Hampshire, United States

REFERENCES:
- [Background] Cleland JA, Fritz JM, Childs JD, Kulig K. Comparison of the effectiveness of three manual physical therapy techniques in a subgroup of patients with low back pain who satisfy a clinical prediction rule: study protocol of a randomized clinical trial [NCT00257998]. BMC Musculoskelet Disord. 2006 Feb 10;7:11. doi: 10.1186/1471-2474-7-11. PMID 16472379